CLINICAL TRIAL: NCT01530841
Title: Prospective Randomized Controlled Single Blind Study of Efficacy and Tolerance of AVAPS Mode Compared to Bilevel Pressure Ventilation un Adult Patients With Myotonic Dystrophy
Brief Title: Efficacy and Tolerance of AVAPS Mode in Myotonic Dystrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Collaborators: Adep Assistance (Other); Philips Respironics (Industry)
Responsible Party: Principal Investigator, david orlikowski, Professor, MD, PhD, Centre d'Investigation Clinique et Technologique 805
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010-A01306-33
Record Dates: First submitted 2012-02-08; First posted 2012-02-10 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Myopathy
Keywords: Myotonic dystrophy type 1; Home ventilation; Respiratory insufficiency; Neuromuscular
MeSH Terms: conditions — Muscular Diseases; Myotonic Dystrophy; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- AVAPS (Experimental): Arm assigned to AVAPS mode for nocturnal ventilation with the same setting than bilevel pressure support but with AVAPS mode activated
  Interventions: Device: Nocturnal ventilation
- Bilevel pressure (Active Comparator): Arm treated only with bilevel pressure support for nocturnal ventilation without activation of AVAPS mode
  Interventions: Device: Nocturnal ventilation

INTERVENTIONS:
Device: Nocturnal ventilation — Home ventilation only the mode AVAPS will be used if the patient is randomized in the experimental group.
  Other Names: BIPAP A30

SUMMARY:
Myotonic dystrophy type 1 is a myopathy with complex respiratory pattern and at risk to develop respiratory failure. Classical mode of ventilation are sometimes not tolerated or ineffective in this population. New modes of nocturnal ventilation by combining both volumetric and barometric advantages. The aim of this study is to compare effect of AVAPS mode to bilevel pressure support.

DETAILED DESCRIPTION:
Justification of study

Respiratory abnormalities are complex in Myotonic dystrophy type 1. Some patients presented with isolated alveolar hypoventilation and breathe rhythm irregularity. Nocturnal ventilation is usually proposed but usual modes of ventilation can't provide enough respiratory assistance for patients especially during REM sleep or too much respiratory assistance increasing the risk of asynchrony. The goal of this study is to evaluate the effect of the mode AVAPS (a mode permitting a pressure support with guaranteed volume and offering advantage of volume and pressure support with Bipap A30 Phillips Respironics) compared to bilevel pressure support.

Main Objective To evaluate efficacy of AVAPS Mode at day 7 on arterial PCO2 under ventilation after launching ventilation.

Secondary Objectives To evaluate efficacy of AVAPS Mode at day 90 on daytime arterial PCO2 after launching ventilation.

To evaluate compliance to ventilation at day 7 and 90. To evaluate clinical efficacy on respiratory symptoms, dyspnea and sleepiness at day 1 and 90.

To evaluate quality of life at day 1 and 90. To evaluate effect of AVAPS on polysomnography, nocturnal SaO2, nocturnal PtCO2.

To evaluate Multiple sleep latency and Maintenance of wakefulness tests at day 90.

To evaluate effect of AVAPS on respiratory parameters VC and mouth maximal pressures.

Type of study: Prospective, monocentre, randomized, controlled single blind study on 2 parallel group.

Number of subjects: 32 patients recruited in home ventilation unit of Raymond Poincaré hospital.

Selection criteria : Patients with Myotonic dystrophy presenting at least one clinical signs : effort or rest dyspnea, orthopnea, sleepiness, morning headache or VC<50% or Pi max< 60 cm H2O or time of SaO2<90% more than 5 minutes and Hypercapnia > 6.0 kPa.

Study process Preceding screening period within the 3 months before inclusion. Day 1 to day 3 baseline evaluation. Day 3 Inclusion and Randomisation Day 3 to 8 Launch of ventilation Day 8 Home discharge Day 90 Evaluation of efficacy (secondary objectives) and observance.

Duration Participation of a patient 3 months. Period of inclusion 24 months. Total duration of study 30 months.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged > 18 years
* Written consent
* DM1 myotonic dystrophy
* One clinical signs dyspnea rest/effort, orthopnea, daytime sleepiness (Epworth> 10), morning headache.

Or restrictive syndrome: VC< 50 % or Pi max <60 cm H2O Or time of nocturnal saturation < 90 %, > 5 minutes. AND Hypercapnia > 6.0 kPa Pregnancy test negative or use of contraception for women in age of procreation

Exclusion Criteria:

* Patient using previously home ventilation within the 6 months before entering the study
* Patient denying home ventilation
* Refusal to sign consent
* impossibility to be followed during 3 months
* Impossibility to apply ventilation at home
* No social/health coverage
* Patient under tutelage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
arterial PCO2 under ventilation | 7 days
  To evaluate efficacy of AVAPS Mode versus bilevel pressure mode at day 7 on arterial PCO2 under ventilation after launching ventilation

SECONDARY OUTCOMES:
daytime arterial PCO2 after launching ventilation. | 90 days
  To evaluate efficacy of AVAPS Mode at day 90 on daytime arterial PCO2 after launching ventilation.
Compliance to ventilation | 7 and 90 days
  To evaluate compliance (h/24h) to ventilation at days 7 and 90.
Symptoms | 90 days
  To evaluate clinical efficacy on respiratory symptoms, dyspnea and sleepiness at day 1 and 90.
Sleep studies | 90 days
  To evaluate effect of AVAPS on polysomnography, nocturnal SaO2, nocturnal PtCO2 at day 90.
OBJECTIVE SLEEPINESS | 90 days
  To evaluate Multiple sleep latency and Maintenance of wakefulness tests at day 90.
Respiratory parameters | 90 days
  To evaluate effect of AVAPS on respiratory parameters VC and mouth maximal pressures.

CONTACTS AND LOCATIONS:
Overall Officials: David ORLIKOWSKI, Md-PhD, Principal Investigator — Raymond Poincare Hospital - Garches - France
Locations (1):
- Home ventilation Unit , Raymond Poincaré hospital, Garches, Paris Area, France